CLINICAL TRIAL: NCT02713867
Title: A Dose Frequency Optimization, Phase IIIB/IV Trial of Nivolumab 240 mg Every 2 Weeks vs Nivolumab 480 mg Every 4 Weeks in Subjects With Advanced or Metastatic Non-small Cell Lung Cancer Who Received up to 12 Months of Nivolumab at 3 mg/kg or 240 mg Every 2 Weeks
Brief Title: A Dose Frequency Optimization,Trial of Nivolumab 240 mg Every 2 Weeks vs Nivolumab 480 mg Every 4 Weeks in Subjects With Advanced or Metastatic Non-small Cell Lung Cancer Who Received Up to 12 Months of Nivolumab at 3 mg/kg or 240 mg Every 2 Weeks
Acronym: CheckMate 384
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CA209-384
Record Dates: First submitted 2016-03-11; First posted 2016-03-21 (Estimated); Results first posted 2020-06-22 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nivolumab 240 mg (Active Comparator): Nivolumab 240 mg Every 2 Weeks
  Interventions: Biological: Nivolumab
- Nivolumab 480 mg (Experimental): Nivolumab 480 mg Every 4 Weeks
  Interventions: Biological: Nivolumab

INTERVENTIONS:
Biological: Nivolumab

SUMMARY:
The primary objective of this study is to compare PFS (progression-free survival) rate at 6 months and at 1 year after randomization, of Nivolumab 480 mg every 4 weeks with nivolumab 240 mg every 2 weeks in subjects with advanced/metastatic (Stage IIIb/IV) NSCLC (non-Sq and Sq).

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Histologically or cytologically documented Squamous or non-Squamous Non-small cell lung cancer (NSCLC) (Stage IIIB/IV), or recurrent or progressive disease following multimodal therapy
* Patients must have received pre-study nivolumab for up to 12 months and have 2 consecutive tumor assessments confirming Complete response (CR), Partial response (PR), or Stable disease (SD)
* Measurable disease before start of pre-study nivolumab treatment
* Eastern Cooperative Oncology Group (ECOG) Performance status (PS) 0-2

Exclusion Criteria:

* Carcinomatous meningitis
* Untreated, symptomatic Central nervous system (CNS) metastases
* Symptomatic interstitial lung disease

Other protocol defined inclusion/exclusion criteria could apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2019-07-15 (Actual); Study Completion 2022-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (129):
- United States (77):
  - Local Institution - 0004, Birmingham, Alabama
  - Local Institution - 0030, Phoenix, Arizona
  - Local Institution - 0041, Phoenix, Arizona
  - CBCC Global Research, Inc., Bakersfield, California
  - Southern California Permanente Medical Group, Bellflower, California
  - St Jude Hospital Yorba Linda, Fullerton, California
  - Local Institution - 0046, Los Angeles, California
  - Local Institution - 0126, Orange, California
  - Torrance Health Association, Redondo Beach, California
  - Sharp Memorial Hospital, San Diego, California
  - Local Institution - 0010, Santa Barbara, California
  - Local Institution - 0044, Santa Maria, California
  - Local Institution - 0130, Vallejo, California
  - Local Institution - 0017, Denver, Colorado
  - Local Institution - 0122, Fort Collins, Colorado
  - Local Institution - 0038, Fort Myers, Florida
  - Local Institution - 0089, Hollywood, Florida
  - Local Institution - 0026, Ocala, Florida
  - Local Institution - 0001, Pensacola, Florida
  - Local Institution - 0039, St. Petersburg, Florida
  - Local Institution - 0008, Athens, Georgia
  - Local Institution - 0142, Columbus, Georgia
  - Local Institution - 0121, Marietta, Georgia
  - Ingalls Health System, Harvey, Illinois
  - Local Institution - 0098, Niles, Illinois
  - Local Institution - 0100, Peoria, Illinois
  - Local Institution - 0143, Urbana, Illinois
  - Local Institution - 0099, Fort Wayne, Indiana
  - Local Institution - 0050, Fort Wayne, Indiana
  - Innova Schar Cancer Institute, Indianapolis, Indiana
  - Local Institution - 0123, Wichita, Kansas
  - Local Institution - 0112, Paducah, Kentucky
  - Mary Bird Perkins Cancer Center, Baton Rouge, Louisiana
  - Local Institution - 0137, New Orleans, Louisiana
  - Local Institution - 0109, Brewer, Maine
  - Local Institution - 0042, Bethesda, Maryland
  - Local Institution - 0125, Springfield, Massachusetts
  - Local Institution - 0136, Southfield, Michigan
  - Local Institution - 0120, Minneapolis, Minnesota
  - Local Institution - 0116, Tupelo, Mississippi
  - Mercy Medical Research Institute, Springfield, Missouri
  - Local Institution - 0014, Omaha, Nebraska
  - Local Institution - 0141, Lebanon, New Hampshire
  - Local Institution - 0035, Albany, New York
  - Local Institution - 0013, Johnson City, New York
  - Local Institution - 0127, Pinehurst, North Carolina
  - Hematology And Oncology Associates, Canton, Ohio
  - Local Institution - 0037, Cincinnati, Ohio
  - Local Institution - 0132, Cincinnati, Ohio
  - MetroHealth Cancer Care Center, Cleveland, Ohio
  - Local Institution - 0129, Massillon, Ohio
  - Hematology Oncology Consultants, Pc, Medford, Oregon
  - Local Institution - 0005, Pittsburgh, Pennsylvania
  - Local Institution - 0020, Charleston, South Carolina
  - Local Institution - 0124, Sioux Falls, South Dakota
  - Jones Clinic PC, Germantown, Tennessee
  - Local Institution - 0036, Nashville, Tennessee
  - Local Institution - 0023, Abilene, Texas
  - Texas Oncology - Amarillo, Amarillo, Texas
  - Local Institution - 0011, Dallas, Texas
  - Local Institution - 0022, Dallas, Texas
  - Texas Oncology, P.A., Denton, Texas
  - Texas Oncology, P.A., El Paso, Texas
  - Local Institution - 0025, Flower Mound, Texas
  - Texas Oncology, P.A., Houston, Texas
  - Texas Oncology, P.A., Longview, Texas
  - Local Institution - 0119, Midland, Texas
  - Texas Oncology, P.A., Plano, Texas
  - Texas Oncology, P.A., San Antonio, Texas
  - Texas Oncology, P.A., Sherman, Texas
  - Texas Oncology, P.A., Sugar Land, Texas
  - Local Institution - 0034, Wichita Falls, Texas
  - Innova Schar Cancer Institute, Falls Church, Virginia
  - Shenandoah Oncology, Winchester, Virginia
  - Cancer Care Northwest, Spokane Valley, Washington
  - Local Institution - 0031, Vancouver, Washington
  - Yakima Valley Memorial Hospital/North Star Lodge, Yakima, Washington
- Australia (10):
  - Local Institution - 0052, St Leonards, New South Wales
  - Local Institution - 0118, Waratah, New South Wales
  - Local Institution - 0117, Westmead, New South Wales
  - Local Institution - 0093, Woolloongabba, Queensland
  - Local Institution - 0054, Bedford Park, South Australia
  - Local Institution - 0056, Elizabeth Vale, South Australia
  - Local Institution - 0055, Kurralta Park, South Australia
  - Local Institution - 0057, Hobart, Tasmania
  - Local Institution - 0053, Heidelberg, Victoria
  - Local Institution - 0058, Murdoch, Western Australia
- Local Institution, Vienna, Austria
- Canada (5):
  - Local Institution - 0059, Newmarket, Ontario
  - Local Institution - 0146, Laval, Quebec
  - Local Institution - 0145, Montreal, Quebec
  - Local Institution, Québec, Quebec
  - Local Institution - 0060, Saint-Jérôme, Quebec
- France (14):
  - Local Institution - 0081, Angers
  - Local Institution - 0105, Angers
  - Local Institution - 0080, Bayonne
  - Local Institution - 0076, Clermont-Ferrand
  - Local Institution - 0077, Le Mans
  - Local Institution - 0072, Mulhouse
  - Local Institution - 0078, Nîmes
  - Local Institution - 0095, Paris
  - Local Institution - 0083, Paris
  - Local Institution, Pontoise
  - Local Institution - 0075, Suresnes
  - Local Institution - 0079, Tours
  - Local Institution - 0097, Vandœuvre-lès-Nancy
  - Local Institution - 0096, Villefranche-sur-Saône
- Germany (14):
  - Local Institution, Bad Berka
  - Local Institution - 0073, Berlin
  - Local Institution - 0063, Dresden
  - Local Institution, Freiburg im Breisgau
  - Local Institution - 0102, Gauting
  - Local Institution - 0062, Greifenstein
  - Local Institution - 0061, Hamburg
  - Local Institution - 0113, Hanover
  - Local Institution - 0064, Kassel
  - Local Institution - 0106, Kiel
  - Local Institution - 0065, Leipzig
  - Local Institution, Lostau
  - Local Institution - 0066, Moers
  - Local Institution - 0067, Nuremberg
- Italy (4):
  - Local Institution - 0086, Localita San Filippo Lucca
  - Local Institution - 0085, Monza
  - Local Institution - 0088, Napoli
  - Local Institution - 0087, Roma
- Spain (4):
  - Local Institution - 0069, Barcelona
  - Local Institution - 0104, El Palmar
  - Local Institution - 0068, Las Palmas de Gran Canaria
  - Local Institution - 0070, Seville

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Nivolumab 480mg: Nivolumab 480mg Q4W
- Nivolumab 240mg: Nivolumab 240mg Q2W
Period: Randomization
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Started (= Participants Randomized) | 180 | 183
Completed (= Participants Treated) | 178 | 180
Not Completed | 2 | 3
Not completed — Other Reason | 2 | 1
Not completed — Participant Withdrew consent | 0 | 2
Period: Treatment Period
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Started (= Started Treatment) | 178 | 180
Completed (= Continuing Treatment Period) | 0 | 0
Not Completed | 178 | 180
Not completed — Other Reasons | 22 | 28
Not completed — Administrative reason by sponsor | 21 | 16
Not completed — No longer meets study criteria | 2 | 1
Not completed — Poor/Non Compliance | 1 | 0
Not completed — Maximum Clinical Benefit | 5 | 6
Not completed — Withdrew consent | 3 | 6
Not completed — Requested to Discontinue | 8 | 8
Not completed — AE unrelated to Study Drug | 11 | 10
Not completed — Death | 7 | 3
Not completed — Study Drug Toxicity | 16 | 19
Not completed — Disease Progression | 82 | 83

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nivolumab 480mg | Nivolumab 240mg | Total
Number analyzed (Participants) | 180 | 183 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 66.4 (9.25) | 66.5 (8.65) | 66.5 (8.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 54 | 103
  Male | 131 | 129 | 260
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 118 | 115 | 233
  Unknown or Not Reported | 59 | 64 | 123
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 7 | 15
  White | 169 | 168 | 337
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 5 | 7

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival Rate (PFSR) at 6 Months
Description: The proportion of participants remaining progression free and surviving at 6 months. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. Note: the appearance of one or more new lesions is also considered progression.
Time Frame: At 6 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of Participants | 0.76 [0.70 to 0.83] | 0.79 [0.73 to 0.85]

2. Primary Outcome: Progression Free Survival Rate (PFSR) at 12 Months
Description: as for outcome 1
Time Frame: At 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of Participants | 0.53 [0.46 to 0.61] | 0.55 [0.47 to 0.62]

3. Secondary Outcome: Progression Free Survival Rate (PFSR) at 24 Months
Description: as for outcome 1
Time Frame: At 24 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of Participants | 0.34 [0.27 to 0.42] | 0.35 [0.28 to 0.43]

4. Secondary Outcome: Progression Free Survival Rate (PFSR) by Tumor Histology at 12 Months
Description: as for outcome 1
Time Frame: At 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of Participants
  Squamous: number analyzed (Participants) | 61 | 64
  Squamous | 0.50 [0.37 to 0.64] | 0.42 [0.29 to 0.55]
  Non Squamous: number analyzed (Participants) | 119 | 119
  Non Squamous | 0.54 [0.45 to 0.63] | 0.60 [0.51 to 0.70]

5. Secondary Outcome: Progression Free Survival Rate (PFSR) by Response Criteria at 12 Months
Description: The proportion of participants remaining progression free and surviving at 12 months. Participants who did not progress or die will be censored on the date of their last evaluable tumor assessment. Progression is defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: At 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of Participants
  Complete Remission (CR)/Partial Remission (PR): number analyzed (Participants) | 61 | 62
  Complete Remission (CR)/Partial Remission (PR) | 0.63 [0.51 to 0.75] | 0.66 [0.53 to 0.78]
  Stable Disease (SD): number analyzed (Participants) | 119 | 121
  Stable Disease (SD) | 0.47 [0.38 to 0.57] | 0.48 [0.39 to 0.58]

6. Secondary Outcome: Overall Survival (OS) Rate at 12 Months
Description: The proportion of participants alive at 12 months. OS is defined as time from the date of randomization to the date of death. Participants who did not die by the end of the study will be censored at the last known date alive.
Time Frame: At 12 Months
Population: All Randomized Participants with a response at 12 months
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 142 | 150
Proportion of participants | 0.851 [0.799 to 0.902] | 0.908 [0.866 to 0.951]

7. Secondary Outcome: Overall Survival (OS) Rate up to 60 Months
Description: The proportion of participants alive up to 60 months. OS is defined as time from the date of randomization to the date of death. Participants who did not die by the end of the study will be censored at the last known date alive.
Time Frame: From randomization to the date of death, Up to 60 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of participants
  12 Months: number analyzed (Participants) | 142 | 150
  12 Months | 0.82 [0.76 to 0.88] | 0.88 [0.83 to 0.93]
  24 Months: number analyzed (Participants) | 104 | 114
  24 Months | 0.62 [0.55 to 0.69] | 0.70 [0.63 to 0.77]
  36 Months: number analyzed (Participants) | 40 | 40
  36 Months | 0.49 [0.42 to 0.57] | 0.57 [0.49 to 0.64]
  48 Months: number analyzed (Participants) | 3 | 2
  48 Months | NA [NA to NA] — Data not calculable due to inability insufficient number of participants for analysis for K-M methodology. | NA [NA to NA] — Data not calculable due to inability insufficient number of participants for analysis for K-M methodology.
  60 Months: number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Overall Survival Rate by Histology at 12 Months
Description: The proportion of participants alive at 12 months. OS is defined as time from the date of randomization to the date of death. Participants who did not die by the end of the study will be censored at the last known date alive.
  OS rate by histology did not have data collected after 12 months randomization.
Time Frame: at 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of participants
  Squamous: number analyzed (Participants) | 61 | 64
  Squamous | 0.74 [0.63 to 0.85] | 0.80 [0.70 to 0.90]
  Non Squamous: number analyzed (Participants) | 119 | 119
  Non Squamous | 0.86 [0.80 to 0.92] | 0.92 [0.87 to 0.97]

9. Secondary Outcome: Overall Survival Rate by Response Criteria at 12 Months
Description: The proportion of participants alive at 12 months. OS is defined as time from the date of randomization to the date of death. Participants who did not die by the end of the study will be censored at the last known date alive.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Stable Disease (SD): Neither sufficient shrinkage from the baseline study to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
  OS rate by response did not have data collected after 12 months randomization.
Time Frame: 12 Months
Population: All Randomized Participants
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 180 | 183
Proportion of participants
  CR/PR: number analyzed (Participants) | 61 | 62
  CR/PR | 0.90 [0.82 to 0.98] | 0.93 [0.87 to 1.00]
  SD: number analyzed (Participants) | 119 | 121
  SD | 0.78 [0.70 to 0.86] | 0.85 [0.78 to 0.92]

10. Secondary Outcome: Percentage of Participants With an Adverse Events (AEs)
Description: Percentage of participants with an Adverse Event due to any cause
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 91.6 | 97.8

11. Secondary Outcome: Percentage of Participants With an Serious Adverse Events (SAEs)
Description: Percentage of participants with an Serious Adverse Event due to any cause.
  A Serious Adverse Event (SAE) is any untoward medical occurrence that at any dose:
  1. results in death
  2. is life-threatening (defined as an event in which the subject was at risk of death at the time of the event; it does not refer to an event which hypothetically might have caused death if it were more severe)
  3. requires inpatient hospitalization or causes prolongation of existing hospitalization
  4. results in persistent or significant disability/incapacity
  5. is a congenital anomaly/birth defect
  6. is an important medical event (defined as a medical event(s) that may not be immediately life-threatening or result in death or hospitalization but, based upon appropriate medical and scientific judgment, may jeopardize the participant or may require intervention [eg, medical, surgical] to prevent one of the other serious outcomes listed in the definition above.)
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 34.8 | 39.4

12. Secondary Outcome: Percentage of Participants With an Adverse Events Leading to Discontinuation (AEsDC)
Description: Percentage of Participants with an Adverse Event leading to discontinuation (AEsDC) due to any cause.
  An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in a clinical investigation participant administered study drug and that does not necessarily have a causal relationship with this treatment.
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 19.1 | 17.8

13. Secondary Outcome: Percentage of Participants With an Immune Mediated Adverse Events (IMAEs)
Description: Percentage of Participants with an Immune Mediated Adverse Events treated with Immune-Modulating Medication
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants
  Diarrhea/Colitis | 3.4 | 5.0
  Hepatitis | 0.0 | 1.7
  Pneumonitis | 3.4 | 3.3
  Nephritis and Renal Dysfunction | 0.6 | 0.0
  Rash | 7.3 | 7.2
  Hypersensitivity/Infusion Reaction | 0.0 | 0.0

14. Secondary Outcome: Percentage of Participants With an Select Adverse Events
Description: Percentage of Participants with an Select Adverse Event due to any cause
  Select adverse events include adverse events in the following systems: Gastrointestinal, Hepatic, Pulmonary, Renal, Skin, Hypersensitivity/Infusion reaction and Endocrine.
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants
  Gastrointestinal | 18.5 | 25.0
  Hepatic | 2.2 | 10.0
  Pulmonary | 6.7 | 5.0
  Renal | 10.1 | 5.6
  Skin | 30.9 | 33.9
  Hypersensitivity/Infusion Reaction | 0.0 | 1.1
  Endocrine | 16.3 | 18.3

15. Secondary Outcome: Percentage of Participants With an Event of Special Interest (ESI)
Description: Other ESI included the following categories: demyelination, encephalitis, Guillain-Barré syndrome (GBS), myasthenic syndrome, pancreatitis, uveitis, myositis, myocarditis, rhabdomyolysis, and Graft Versus Host Disease (GVHD).
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants
  Pancreatitis | 1.1 | 2.8
  demyelination | 0 | 0
  encephalitis | 0 | 0
  GBS | 0 | 0
  myasthenic syndrome | 0 | 0
  uveitis | 0 | 0
  myositis | 0 | 0
  myocarditis | 0 | 0
  rhabdomyolysis | 0 | 0
  GVHD | 0 | 0

16. Secondary Outcome: Percentage of Participants Who Experienced Death
Description: Percentage of Participants who experienced Death due to any cause
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Percentage of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Percentage of Participants | 49.4 | 43.9

17. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities
Description: Number of participants with any laboratory test result that is clinically significant or meets the definition of an SAE (Grade 3+4 combined)
Time Frame: Between first dose and 100 days after last dose of study therapy (Approximately Up to 16 months)
Population: All Treated Participants
Measure: Number; unit: Number of Participants
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
Number analyzed (Participants) | 178 | 180
Number of Participants
  Alanine Aminotransferase | 1 | 1
  Alkaline Phosphate | 1 | 0
  Aspartate Aminotransferase | 1 | 2
  Bilirubin, Total | 1 | 1
  Creatinine | 1 | 2
  Hemoglobin | 0 | 4
  Hypercalcemia | 2 | 5
  Hyperkalemia | 4 | 3
  Hypermagnesemia | 4 | 5
  Hypernatremia | 0 | 0
  Hypocalcemia | 4 | 6
  Hypokalemia | 3 | 6
  Hypomagnesemia | 3 | 2
  Hypnatremia | 6 | 7
  Leukocytes | 1 | 3
  Lymphocytes | 22 | 21
  Neutrophils | 3 | 4
  Platelet Count | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse events and SAEs: between first dose and 100 days after last dose of study therapy (On average of 16 months up to a maximum of 56 months). All Cause Mortality, from randomization to study completion.: Approximately 5 years and 8 months.
Description: The number at Risk for All-Cause Mortality represents all Randomized Participants to study completion.
  The number at Risk for Serious Adverse Events and Other (Not Including Serious) Adverse Events represents all participants that received at least 1 dose of study medication" or similar.
Arm/Group | Nivolumab 480mg | Nivolumab 240mg
All-Cause Mortality (participants affected / at risk) | 88/180 | 79/183
Serious Adverse Events (participants affected / at risk) | 62/178 | 71/180
Other Adverse Events (participants affected / at risk) | 141/178 | 168/180
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 480mg (N=178) | Nivolumab 240mg (N=180)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Coronary artery occlusion (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 2
Supraventricular tachycardia (Cardiac disorders) | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 1 | 0
Hypophysitis (Endocrine disorders) | 1 | 0
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Autoimmune colitis (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 4 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal pain (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Drowning (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Sudden death (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 2
Lung abscess (Infections and infestations) | 0 | 1
Medical device site cellulitis (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 9
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia pneumococcal (Infections and infestations) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection bacterial (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Urosepsis (Infections and infestations) | 1 | 0
Animal bite (Injury, poisoning and procedural complications) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haematuria (Injury, poisoning and procedural complications) | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 2
Wound evisceration (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1
Soft tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 | 1
Thoracic spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Glottis carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Laryngeal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 9
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Rectal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery occlusion (Nervous system disorders) | 0 | 1
Cerebral ischaemia (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 1
Nystagmus (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 2
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 0 | 1
Subcapsular renal haematoma (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Aortic aneurysm (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 1
Peripheral artery occlusion (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Nivolumab 480mg (N=178) | Nivolumab 240mg (N=180)
Anaemia (Blood and lymphatic system disorders) | 11 | 19
Hypothyroidism (Endocrine disorders) | 21 | 17
Abdominal pain (Gastrointestinal disorders) | 10 | 7
Abdominal pain upper (Gastrointestinal disorders) | 5 | 10
Constipation (Gastrointestinal disorders) | 19 | 22
Diarrhoea (Gastrointestinal disorders) | 30 | 41
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 7 | 11
Nausea (Gastrointestinal disorders) | 12 | 29
Vomiting (Gastrointestinal disorders) | 12 | 20
Asthenia (General disorders) | 24 | 24
Fatigue (General disorders) | 28 | 40
Non-cardiac chest pain (General disorders) | 5 | 10
Oedema peripheral (General disorders) | 11 | 15
Pyrexia (General disorders) | 14 | 14
Bronchitis (Infections and infestations) | 17 | 23
Nasopharyngitis (Infections and infestations) | 11 | 16
Pneumonia (Infections and infestations) | 8 | 10
Rhinitis (Infections and infestations) | 0 | 10
Sinusitis (Infections and infestations) | 7 | 10
Upper respiratory tract infection (Infections and infestations) | 10 | 16
Urinary tract infection (Infections and infestations) | 5 | 11
Fall (Injury, poisoning and procedural complications) | 8 | 10
Alanine aminotransferase increased (Investigations) | 2 | 9
Amylase increased (Investigations) | 5 | 9
Aspartate aminotransferase increased (Investigations) | 1 | 9
Blood creatinine increased (Investigations) | 14 | 7
Lipase increased (Investigations) | 8 | 14
Weight decreased (Investigations) | 8 | 20
Decreased appetite (Metabolism and nutrition disorders) | 15 | 20
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 9
Hyperkalaemia (Metabolism and nutrition disorders) | 4 | 15
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 9
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 10
Hypophosphataemia (Metabolism and nutrition disorders) | 3 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 24 | 37
Back pain (Musculoskeletal and connective tissue disorders) | 24 | 19
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 11
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 15
Dizziness (Nervous system disorders) | 5 | 17
Headache (Nervous system disorders) | 14 | 15
Insomnia (Psychiatric disorders) | 6 | 20
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 12
Cough (Respiratory, thoracic and mediastinal disorders) | 23 | 36
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 26
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 10 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 12
Pruritus (Skin and subcutaneous tissue disorders) | 30 | 42
Rash (Skin and subcutaneous tissue disorders) | 10 | 9
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 10 | 6
Hypertension (Vascular disorders) | 10 | 12

LIMITATIONS AND CAVEATS:
No formal statistical analyses were conducted. Median OS was not reached in either arm.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-06-26): https://cdn.clinicaltrials.gov/large-docs/67/NCT02713867/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-28): https://cdn.clinicaltrials.gov/large-docs/67/NCT02713867/SAP_000.pdf